CLINICAL TRIAL: NCT02321267
Title: Cohort Study of the Clinical Course of Macular Diseases in Kagawa (Kagawa Macula Cohort Study)
Brief Title: Cohort Study of the Clinical Course of Macular Diseases in Kagawa
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kagawa University (Other)
Responsible Party: Principal Investigator, Akitaka Tsujikawa, Professor and Chairman, Kagawa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H26-035
Record Dates: First submitted 2014-12-10; First posted 2014-12-22 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Macular Disease
Keywords: AMD; PCV; RAP; RVO; DME; ERM; MH; mCNV
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; aflibercept; pegaptanib; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macular disease with adequate treatments (Other): Macular diseases can be treated with most appropriate treatment, including pegaptanib, ranibizumab, afibercept, visudyne, or vitrectomy.
  Interventions: Drug: ranibizumab, aflibercept, pegaptanib, verteporphin

INTERVENTIONS:
Drug: ranibizumab, aflibercept, pegaptanib, verteporphin — ranibizumab, intravitreal injections, 0.5mg, monthly or less aflibercept,intravitreal injections, 2.0mg, monthly or less pegaptanib, intravitreal injections, 0.3mg, every 6-week pars plana vitrectomy, once verteporphin, iv, 6mg/㎡
  Other Names: Lucentis, Eylea, Macugen, Vizudyne

SUMMARY:
Macular diseases often cases severe visual impairment. Recent clinical introduction of anti-vascular endothelial growth factor agents may change the clinical course of various macular diseases, including age-related macular degeneration (AMD), polypoidal choroidal vasculopathy (PCV), retinal angiomatous proliferation (RAP), central serous chorioretinopathy (CSC), myopic choroidal neovascularization (CNV), retinal vein occlusion (RVO), diabetic macular edema (DME), and so forth. The advance in vitrectomy improve visual outcomes in some maculae diseases, including epiretinal membrane (ERM), macular hole (MH), vitreomacular traction syndrome (VMTS).

Patients with such macular diseases are registered and are followed up for 5 years with appropriate treatment for each patient. By the analysis of the correlation between initial examinations and final visual acuity, factors associated with good visual prognosis will be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit Department of Ophthalmology, Kagawa University Hospital with macular diseases, such as AMD, PCV, RAP, RVO, DME, ERM, MH, VMTS.
* Patients who are agreed with the participation of this study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-12; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of best-collected visual acuity from baseline at 5 years | Five years after the registration

CONTACTS AND LOCATIONS:
Overall Officials: Akiataka Tsujikawa, MD, Principal Investigator — Kagawa Univerisity Faculty of Medicine
Locations (1):
- Kagawa University Faculty of Medicine, Hiragi, Kagawa-ken, Japan